CLINICAL TRIAL: NCT00030277
Title: Feasibility Study for Locally Recurrent Prostate Cancer Treatment With HIFU Using the SONABLATE System
Brief Title: High-Intensity Focused Ultrasound in Treating Patients With Locally Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Focus Surgery (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: FOCUS-G000280; CDR0000069125 (Registry Identifier: PDQ (Physician Data Query)); IUMC-010235; NCI-V01-1683
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-12

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation

INTERVENTIONS:
Procedure: high-intensity focused ultrasound ablation

SUMMARY:
RATIONALE: Highly focused ultrasound energy may be able to kill cancer cells by heating the tumor without affecting the surrounding tissue.

PURPOSE: This phase I trial is studying focused ultrasound energy to see how well it works in treating patients with locally recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of Sonablate to focus ultrasound waves for the purpose of selectively destroying prostate cancer tissue, with resultant drop in PSA levels to below 0.5 ng/mL and negative biopsy for cancer cells, in patients with locally recurrent prostate cancer.

OUTLINE: Patients are stratified according to prior treatment failure (brachytherapy vs post-external beam radiotherapy).

A probe is inserted into the rectum. High-intensity focused ultrasound (HIFU) energy using the Sonablate system is delivered to the prostate tissue over approximately 2 hours. Patients with residual cancer lesion (by biopsy), PSA greater than 0.5 ng/mL or increasing PSA levels taken 2 months apart, visible prostate tissue on ultrasound, and no local or distant metastases after day 90 undergo retreatment with HIFU.

Patients are followed at 2, 14, 30, 90, and 180 days.

PROJECTED ACCRUAL: A total of 20 patients (10 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally recurrent prostate cancer after prior brachytherapy or external-beam radiotherapy for initial diagnosis of organ-confined disease (clinical stage T1 or T2 only)

  * Prostatic fossa biopsy positive for cancer cells
* Gleason score no greater than 7
* PSA levels 0.5-10 ng/mL
* Able to adequately visualize local recurrence on transrectal ultrasound imaging
* No prostate calcification greater than 5 mm
* No metastases by bone scan

PATIENT CHARACTERISTICS:

Age:

* 40 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No bleeding disorder as determined by abnormal PT and PTT

Renal:

* No active urinary tract infection
* No history of urinary bladder neck contracture

Other:

* No prior allergy to latex
* No Anesthesia Surgical Assignment (ASA) category IV or greater
* No interest in future fertility
* No history of inflammatory bowel disease
* No other concurrent major nonmalignant debilitating illness
* No other prior or concurrent malignancy except skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for prostate cancer

Chemotherapy:

* No prior chemotherapy for prostate cancer

Endocrine therapy:

* At least 3 months since prior hormonal therapy (including finasteride) for prostate cancer

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* No prior radical prostatectomy
* No prior transurethral resection of prostate
* No prior urethral stent
* No prior major rectal surgery

Other:

* No prior thermotherapy
* No other prior therapy for prostate cancer
* No concurrent warfarin or other anticoagulant

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2001-10; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael O. Koch, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Long Island College Hospital, Brooklyn, New York